CLINICAL TRIAL: NCT01354899
Title: A Multi-Centre, Post CE Mark, Open Study to Evaluate the Performance of Thin Self-adherent Dressing Coated With a Soft Silicone Layer on Subjects With a High Risk of Skin Breakdown
Brief Title: A Open Study to Evaluate the Performance of Dressing on Subject With High Risk of Skin Breakdown
Status: Completed | Type: Observational
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Other Study IDs: WINDOW 01; Window 02
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The rational for the study is to add a thin self-adherent dressing on critically ill patients. Evaluate if the dressing might protect the skin for further breakdown.Participants will be followed for the duration of hospital stay, an expected average of 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Braden total score ≤ 12 at enrolment
* Male or female, ≥ 18 at enrolment
* No skin- breakdown
* Subject or family member is able to understand and comply with the requirements of the study, judged by the investigator

Exclusion Criteria:

* Risk area dosen´t fit the dressing size
* Documented skin disease
* Kown allergy to any of the components in the dressing
* Previous enroled in present study
* Subject included in other ongoing clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients at ICU.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Faergemann, Professor, Principal Investigator — Dermatology Department Sahlgrenska University Gothenburg
Locations (1):
- Dermatology Department, Gothenburg, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from 17 May 2011 - 29 June 2011. The study was conducted at four intensive care units in Sweden.
Pre-assignment Details: There was no wash-out or run-in phase included in the study.
Groups:
- Window: WindowTM is a protective layer that may reduce the shear and friction on the skin and may help to prevent skin breakdown. Window TM provides instant tack adhesion that minimizes the requirement of extra pressure in order to fixate well. The product does not leave residues and the adhesion level does not increase over time.
  Critically ill subjects treated within intensive care have a high risk to developing pressure ulcers, this is because they are almost invariably limited in their overall physical activity changing their position in bed and it is very common with impaired circulation and/or using specific medication which also can lead to high risk of developing pressure ulcer.
Period: Overall Study
Arm/Group | Window
Started | 24
Completed | 21
Not Completed | 3
Not completed — discharge from the hospital | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Window
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Region of Enrollment [Number; unit: participants]
  Sweden | 24

OUTCOME MEASURES:

1. Primary Outcome: Erythema (No/Yes)
Description: Measure number of skin breakdown during from enrolment to termination.
Time Frame: During 5 days
Measure: Number; unit: participants
Arm/Group | Window
Number analyzed (Participants) | 24
participants
  No | 21
  Yes | 3

2. Secondary Outcome: Overall Experience of Use of the Dressing
Description: Overall experience of use of the dressing rated on a scale from Very Poor, Poor, Good, Very Good, Excellent
Time Frame: During 5 days
Measure: Number; unit: participants
Arm/Group | Window
Number analyzed (Participants) | 24
participants
  Very poor | 1
  Poor | 3
  Good | 10
  Very good | 9
  Excellent | 1

ADVERSE EVENTS:
Time Frame: Adverse Event were collected from enrollment to termination ( 5 days)
Arm/Group | Window
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 7/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Window (N=24)
Death (Vascular disorders) | 1 (1) — Serious medical condition with multiple organ failure after acute abdominal aortic aneurysm rupture with a bleeding of 28000ml. The patient condition deteriorated despite intensive care treatment with ventilator, dialysis and vasopressor drugs.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Window (N=24)
Brady cardia (Cardiac disorders) | 1 (1)
Pressure Ulcer (Skin and subcutaneous tissue disorders) | 4 (5)
Pneumoni (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachy Cardia (Cardiac disorders) | 1 (1)
Arterial Flutter (Cardiac disorders) | 1 (1)
Thromboflebitis in right arm (Infections and infestations) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No